CLINICAL TRIAL: NCT00347620
Title: Improving Vision and Quality of Life in the Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Retirement Research Foundation (Other); National Institute on Aging (NIA) (NIH); National Eye Institute (NEI) (NIH); Research to Prevent Blindness (Other); EyeSight Foundation of Alabama (Other); Pearle Vision Foundation (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000-072
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-03

CONDITIONS: Refractive Error; Cataract
MeSH Terms: conditions — Refractive Errors; Cataract | interventions — Eyeglasses; Cataract Extraction

INTERVENTIONS:
Device: spectacles
Procedure: Cataract Surgery

SUMMARY:
The primary purpose of this study is to evaluate whether interventions to improve vision in nursing home residents have an impact on residents' health-related quality of life. The interventions being evaluated are correction of refractive error (near-sightedness, far-sightedness, presbyopia) and cataract surgery.

DETAILED DESCRIPTION:
The purpose of this project is two-fold: 1.) to establish the psychometric properties of the Nursing Home Vision-Specific Health-Related Quality of Life (HRQOL) instrument, and; 2.) to evaluate the responsiveness of this instrument. Responsiveness will be assessed in two independent preliminary prospective intervention evaluations. The first responsiveness evaluation will involve a new spectacle intervention and the second will involve first eye cataract surgery. In addition, we will examine the association between the responsiveness of this instrument, and changes in visual functioning measures and other demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* at least 60 years of age or older
* expected to stay in facility foe at least 8 months
* stable medical condition
* moderately cognitively impaired or better

Exclusion Criteria:

* those not meeting inclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2000-08; Study Completion 2003-12

PRIMARY OUTCOMES:
vision-targeted health-related quality of life

SECONDARY OUTCOMES:
depression
generic health-related quality of life
functional independence
participation in group activities
physical activities
falls
life space

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owsley, PhD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (17):
- United States (17):
  - Integrated Health Services at Briarcliff, Alabaster, Alabama
  - Shelby Ridge Nursing Home, Alabaster, Alabama
  - Livingston Health Care Center, Bessemer, Alabama
  - Southgate Village, Bessemer, Alabama
  - Beverly Healthcare Meadowood, Bessemer, Alabama
  - Fair Haven Retirement Center, Birmingham, Alabama
  - Beverly Healthcare Center Forestdale, Birmingham, Alabama
  - Beverly Healthcare East, Birmingham, Alabama
  - South Haven, Birmingham, Alabama
  - Fairview Health & Rehabilitation Center, Birmingham, Alabama
  - Estes Nursing Facility Civic Center, Birmingham, Alabama
  - Estes Nursing Facility Northway, Birmingham, Alabama
  - Beverly Healthcare Riverchase, Birmingham, Alabama
  - Beverly Health Care Center West, Fairfield, Alabama
  - The Self Nursing Home, Inc, Hueytown, Alabama
  - Beverly Healthcare Pleasant Grove, Pleasant Grove, Alabama
  - Consult America Cottage Hills, Pleasant Grove, Alabama

REFERENCES:
- [Derived] Owsley C, McGwin G Jr, Scilley K, Meek GC, Seker D, Dyer A. Effect of refractive error correction on health-related quality of life and depression in older nursing home residents. Arch Ophthalmol. 2007 Nov;125(11):1471-7. doi: 10.1001/archopht.125.11.1471. PMID 17998508